CLINICAL TRIAL: NCT01934361
Title: Phase Ib/II Multicenter Study of Buparlisib Plus Carboplatin or Lomustine in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Phase Ib/II Study of Buparlisib Plus Carboplatin or Lomustine in Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120E2102; 2013-003129-27 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2013-09-04 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: BKM120; Recurrent glioblastoma multiforme; rGBM; buparlisib
MeSH Terms: conditions — Glioblastoma | interventions — NVP-BKM120; Carboplatin; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lomustine+ buparlisib (Phase Ib) (Experimental)
  Interventions: Drug: buparlisib; Drug: lomustine
- carboplatin+ buparlisib (Phase Ib) (Experimental)
  Interventions: Drug: buparlisib; Drug: carboplatin
- lomustine+ buparlisib (Phase II) (Experimental)
  Interventions: Drug: buparlisib; Drug: lomustine
- lumustine + placebo (Phase II) (Placebo Comparator)
  Interventions: Drug: lomustine; Drug: placebo
- carboplatin+ buparlisib (Phase II) (Experimental)
  Interventions: Drug: buparlisib; Drug: carboplatin

INTERVENTIONS:
Drug: buparlisib — Buparlisib administered orally on a continuous daily schedule. Buparlisib is manufactured as 10mg and 50mg hard gelatin capsules.
  Arms: Lomustine+ buparlisib (Phase Ib); carboplatin+ buparlisib (Phase II); carboplatin+ buparlisib (Phase Ib); lomustine+ buparlisib (Phase II)
Drug: carboplatin — Carboplatin intravenous infusion will be administered at a dose of AUC 5 in a 21 day cycle (every 3 weeks).
  Arms: carboplatin+ buparlisib (Phase II); carboplatin+ buparlisib (Phase Ib)
Drug: lomustine — Lomustine will be administered as a single oral dose of 100 mg/m² every 6 weeks in a 42 day cycles.
  Arms: Lomustine+ buparlisib (Phase Ib); lomustine+ buparlisib (Phase II); lumustine + placebo (Phase II)
Drug: placebo — Placebo will be administered orally on a continuous QD dosing schedule for cycles of 42 days. Buparlisib matching placebo is manufactured as 10 mg and 50 mg hard gelatin capsules.
  Arms: lumustine + placebo (Phase II)

SUMMARY:
This is a multi-center, phase Ib/ II study (two parts) with patients that had recurrent glioblastoma multiforme. The first part (phase Ib) was to investigate the maximum tolerated dose/Recommended phase ll dose (MTD/RP2D) of once daily buparlisib in combination with every-three-week carboplatin or buparlisib once daily in combination with every-six-week lomustine (CCNU) using a Bayesian model. Once MTD/ RP2D is established in either of the 2 arms, the corresponding phase II portion of the study was to start. Phase II was to assess the treatment effect of buparlisib in combination with carboplatin in terms of Progression Free Survival (PFS) and was to compare the treatment effect of buparlisib with lomustine versus lomustine plus placebo in terms of PFS.

A preliminary assessment for both combinations (buparlisib plus carboplatin or lomustine) demonstrated that there was not enough antitumor activity compared to historical data with single agent carboplatin or lomustine. Based on the overall safety profile, and preliminary anti-tumor activity observed in this study, Novartis decided that no additional patients would be enrolled into this study. As a consequence, the Phase II part of the study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult ≥ 18 years old at the time of informed consent.
* Patient has histologically confirmed diagnosis of GBM with documented recurrence after first line treatment including radiotherapy and TMZ (SoC), not suitable for curative surgery or re-irradiation.
* Patient has at least one measurable and/or non-measurable lesion as per RANO criteria
* Patient has recovered (to Grade ≤1) from all clinically significant toxicities related to prior antineoplastic therapies.
* Patient has Karnofsky performance status (KPS) ≥70%.
* Patient has adequate organ and bone marrow functions:

  * Absolute Neutrophils Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L (in case of transfusion stable for ≥14 days prior to treatment start)
  * Hemoglobin ≥ 9.0 g/dL (in case of transfusion stable for ≥14 days prior to treatment start)
  * INR ≤ 1,5
  * Serum Creatinine ≤ 1.5 x ULN, or Creatinine Clearance > 45mL/min
  * Potassium and calcium (corrected for albumin), sodium and magnesium within institutional normal limits
  * Serum Bilirubin ≤ ULN, AST and ALT ≤ ULN
  * HbA1c ≤ 8%
  * Fasting plasma glucose (FPG) ≤ 120 mg/dL or ≤ 6.7 mmol/L
* Patient has tumor tissues available (archival or fresh).

Exclusion Criteria:

* Patient has received previous treatment with PI3K inhibitors, lomustine or carboplatin.
* Patient has received previous antineoplastic treatment for recurrent GBM (e.g. VEGF inhibitors, cytotoxic agents).
* Patient has received more than one line of cytotoxic chemotherapy
* Patient has concurrent use of anti-neoplastic agents including investigational therapy
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed.
* Patient is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated. Switching to a different medication prior to randomization is allowed.
* Patient is currently receiving an enzyme-inducing anti-epileptic drug (EIAED). The patient must have discontinued EIAED therapy for at least two weeks prior to starting study drug.

Other protocol-defined Inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Number of Total Dose-limiting Toxicity (DLT) during Dose Escalation part to determine Maximum Tolerated Dose (MTD) [Phase Ib] | Cycle 1 (21 days carboplatin combination or 42 days lomustine combination )
  Maximum Tolerated Dose (MTD) is defined as the highest BKM120 dosage that does not cause medically unacceptable Dose Limiting Toxicities (DLTs) in more than 35% of the treated patients during the first cycle of treatment. DLT is defined as treatment-related toxicity occurring during the phase Ib cycle 1 and meeting specific protocol-predefined criteria. The information will be integrated in a Bayesian logistic regression model with overdose control to estimate the MTD.
12 week Progression Free Survival (PFS) rate (Phase II- Carboplatin combination) | 12 weeks
  12-week Progression Free Survival (PFS) is defined as the percentage of patients who are progression free 12 weeks after the date of the start of the treatment ("success"). Patients who progressed, died or discontinued within the 12 weeks of observation are counted as "failure".
Progression Free Survival (PFS) [phase II lomustine combinations] | Randomization until date of the event (expected average 3 months).
  Progression Free Survival (PFS) is defined as the time from date of randomization to the date of the event, which is the first radiologically documented disease progression [per local investigator assessment according to Response Assessment in Neuro-Oncology (RANO) criteria] or death due to any cause.

SECONDARY OUTCOMES:
Frequency and severity of Adverse Events (AEs) [Phase Ib, Phase II, all treatment arms] | Until 30 days after treatment discontinuation
  The incidence of Adverse Events (AEs) summarized by system organ class and or preferred term, severity (based on Common Terminology Criteria for Adverse Events (CTCAE) grades version 4), type of AE, relation to study treatment.
Overall Response Rate (ORR) as per Response Assessment in Neuro-Oncology (RANO) [Phase Ib , both combinations] | Baseline, every 6 weeks from treatment start until disease progression or until start of another antineoplastic treatment or death which ever occurs first up to 1 year
  Overall response rate (ORR) is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), based on the investigator assessment as per Response Assessment in Neuro-Oncology (RANO) criteria.
Progression Free Survival (PFS) [Phase Ib- both combinations] | Time from treatment start to the date of the event (expected average 3 months)
  Progression Free Survival (PFS) is defined as time from date of treatment start to the date of the event, which is the first radiologically documented disease progression or death due to any cause per local investigator assessment.
Overall response rate (ORR) [Phae II, carboplatin combination] | Baseline, every 6 weeks from treatment start until disease progression or until start of another antineoplastic treatment or death which ever occurs first up to 1 year
  Overall response rate (ORR) is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), based on the investigator assessment as per Response Assessment in Neuro-Oncology (RANO) criteria.
Progression Free Survival (PFS) [Phase II, carboplatin combination] | Time from treatment start to the date of the event (Expected average: 3 months)
  Progression Free Survival (PFS) is defined as time from date of treatment start to the date of the event, which is the first radiologically documented disease progression or death due to any cause per local investigator assessment.
24 week Progression Free Survival (PFS) rate (Phase II carboplatin combination) | 24 weeks
  24 weeks Progression Free Survival (PFS) is defined as the percentage of patients who are progression free 24 weeks after the date of the start of the treatment ("success"). Patients who progressed, died or discontinued within the 24 weeks of observation are counted as "failure".
Overall Survival (OS) (Phase II Carboplatin combination) | 12 months
  Overall survival (OS) is defined as the time from the date of randomization for buparlisib + lomustine / placebo + lomustine Phase II, or the time from the first study drug intake for buparlisib + carboplatin Phase II, to the date of death due to any cause.
Overall Response Rate (ORR) (Phase II Lomustine combinations) | Baseline, every 6 weeks from treatment start until disease progression or until start of another antineoplastic treatment or death which ever occurs first up to 1 year
  Overall response rate (ORR) is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), based on the investigator assessment as per Response Assessment in Neuro-Oncology (RANO) criteria.
12 week Progression Free Survival (PFS) rate (Phase II- lomustine combinations) | 12 weeks
  12-week Progression Free Survival (PFS) is defined as the percentage of patients who are progression free 12 weeks after the date of the start of the treatment ("success"). Patients who progressed, died or discontinued within the 12 weeks of observation are counted as "failure".
24 week Progression Free Survival (PFS) rate (Phase II- lomustine combinations) | 24 weeks
  24 weeks Progression Free Survival (PFS) is defined as the percentage of patients who are progression free 24 weeks after the date of the start of the treatment ("success"). Patients who progressed, died or discontinued within the 24 weeks of observation are counted as "failure".
Overall survival (OS) [Phase II lomustine combinations] | 12 months
  Overall survival (OS) is defined as the time from the date of randomization for buparlisib + lomustine / placebo + lomustine Phase II, or the time from the first study drug intake for buparlisib + carboplatin Phase II, to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (5):
  - Barrow Neurological Insitute St. Joseph's Hospital, Phoenix, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenthal M, Clement PM, Campone M, Gil-Gil MJ, DeGroot J, Chinot O, Idbaih A, Gan H, Raizer J, Wen PY, Pineda E, Donnet V, Mills D, El-Hashimy M, Mason W. Buparlisib plus carboplatin or lomustine in patients with recurrent glioblastoma: a phase Ib/II, open-label, multicentre, randomised study. ESMO Open. 2020 Jul;5(4):e000672. doi: 10.1136/esmoopen-2020-000672. PMID 32665311
- See also: Results for CBMK120E2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16410